CLINICAL TRIAL: NCT01742065
Title: Strategies and Opportunities to Stop Colon Cancer in Priority Populations
Acronym: STOPCRC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: UH3CA188640 (NIH); 1UH2AT007782-01 (NIH)
Record Dates: First submitted 2012-12-03; First posted 2012-12-05 (Estimated); Results first posted 2019-04-23 (Actual); Last update posted 2019-04-23 (Actual); Status verified 2019-04

CONDITIONS: Colorectal Cancer
Keywords: Colorectal Cancer Screening; Cancer Screening; Pragmatic Trial
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (No Intervention): Clinics in usual care will go about clinic practices to complete recommended screening for colorectal cancer.
- Auto Plus (Active Comparator): Clinics randomized to the Auto-Plus arm will engage in all activities (send an introductory letter to participants, then a FIT Kit, then a reminder letter encouraging the return of the FIT Kit) in addition to a PDSA (Plan Do Study Act) cycle to refine or improve their process.
  Interventions: Other: Auto Plus

INTERVENTIONS:
Other: Auto Plus — Clinics randomized to the Auto-Plus arm will engage in all activities in the Auto arm (send an introductory letter to participants, then a FIT Kit, then a reminder letter encouraging the return of the FIT Kit) in addition to one other outreach effort.
  Arms: Auto Plus

SUMMARY:
Only an estimated 50 million US adults aged 50-75 are up-to-date on colorectal cancer (CRC) screening according to guidelines set by the federal government. CRC is 90% curable with timely detection and appropriate treatment of precancerous polyps; increased screening could reduce incidence by up to 50%. Groups least likely to undergo screening, those with minimal education, low income, low access to health care, recent immigrants or Hispanics, are the same people who frequently receive care at Federally Qualified Healthcare Center's (FQHCs). The use of fecal occult blood tests (FOBT) and fecal immunochemical tests (FIT) is exceedingly low in FQHCs (7-9% of patients in the past year) and far below national averages and target rates. Our results will provide valuable information on how to use electronic health record (EHR) resources to optimize guideline-based screening in FQHC clinics whose patient populations have disproportionately low CRC screening rates.

This project, in conjunction with the research team, will use an advisory panel to direct the research activities. The advisory panel will be made up of clinicians, leaders, researchers, and patients. The panel and team will guide the development of materials, the outreach to patients, and the research protocol to best reach FQHC patients who are due for colorectal cancer screening.

This project will be conducted in two phases, Phase I is conducting a pilot at two FQHC's, and Phase II is rolling out the intervention to between 20-30 clinics.

DETAILED DESCRIPTION:
Phase I (Pilot Aims)

* Aim 1 Conduct preliminary analyses of EHR data at two pilot clinics.
* Aim 2: Use codes and methods developed in Aim 1 to test the feasibility, reach, effectiveness, and cost of an EHR-based CRC screening intervention using a subset of 100 patients at each of two pilot clinics. We will use codes defined in Aim 1 to create a Solutions-based, Epic-integrated system to track CRC screening, mail FIT kits, and track patient test results and receipt of follow-up care. The system will be pilot-tested in two clinics.
* Aim 3: Use results from the pilot intervention to prepare for a large-scale, cluster-randomized pragmatic trial across 18 OCHIN clinics (see Phase II).

Transition from Phase I to Phase II

-Changes to our original proposal include going from a three arm to a two-arm pragmatic cluster trial with revised evaluation and power calculation and refinements to the intervention components for both usual care (now described as enhanced usual care) and the intervention (now described as enhanced auto).

Phase II (Full trial Aims)

* Primary Aim 1. Assess the effectiveness of a large-scale, two-arm CRC screening program among diverse CLINIC patients, and assess difference in CRC screening outcomes (overall and by age, sex, insurance status, Hispanic ethnicity/race). The intervention will consist of an automated data-driven, EHR-linked program for mailing FIT kits (with linguistically appropriate pictographic instructions and return postage) to patients due for CRC screening.
* Primary Aim 2. Assess the costs and long-term cost-effectiveness of the automated program.

We have also included two secondary aims:

* Secondary Aim 1. Assess adoption, implementation, reach and potential maintenance and spread of the program, using a mixed-method rapid assessment process, field notes, and other ethnographic data.
* Secondary Aim 2. Adapt and pilot-test the adaptation of STOP CRC in an alternate EHR platform, Allscripts, and develop an implementation guide to assist sites in adopting the program.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 50-74 with no evidence of a colonoscopy within 9 years or fecal testing within 11 months, and no history of colorectal disease will be eligible to receive a mailed FIT.

Exclusion Criteria:

* End Stage Renal Disease (ESRD)
* Hospice/Nursing Home

Ages: 50 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62155 (Actual)
Dates: Start 2013-01; Primary Completion 2016-02 (Actual); Study Completion 2018-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gloria Coronado, PhD, Principal Investigator — The Center for Health Research, Kaiser Permanente Northwest; Beverly Green, PhD, Principal Investigator — Kaiser Permanente
Locations (8):
- United States (8):
  - Open Door Health Center, Arcata, California
  - Mosaic Medical, Bend, Oregon
  - Benton and Linn County Health Centers, Corvallis, Oregon
  - Virginia Garcia Memorial Health Center, Hillsboro, Oregon
  - La Clinica Health Care, Medford, Oregon
  - Community Health Center, Medford, Oregon
  - Multnomah County Health Department, Portland, Oregon
  - Oregon Health and Science University, Scappoose, Oregon

REFERENCES:
- [Background] Coronado GD, Sanchez J, Petrik A, Kapka T, DeVoe J, Green B. Advantages of wordless instructions on how to complete a fecal immunochemical test: lessons from patient advisory council members of a federally qualified health center. J Cancer Educ. 2014 Mar;29(1):86-90. doi: 10.1007/s13187-013-0551-4. PMID 24057692
- [Background] Coronado GD, Vollmer WM, Petrik A, Taplin SH, Burdick TE, Meenan RT, Green BB. Strategies and Opportunities to STOP Colon Cancer in Priority Populations: design of a cluster-randomized pragmatic trial. Contemp Clin Trials. 2014 Jul;38(2):344-9. doi: 10.1016/j.cct.2014.06.006. Epub 2014 Jun 14. PMID 24937017
- [Background] Coronado GD, Vollmer WM, Petrik A, Aguirre J, Kapka T, Devoe J, Puro J, Miers T, Lembach J, Turner A, Sanchez J, Retecki S, Nelson C, Green B. Strategies and opportunities to STOP colon cancer in priority populations: pragmatic pilot study design and outcomes. BMC Cancer. 2014 Feb 26;14:55. doi: 10.1186/1471-2407-14-55. PMID 24571550
- [Background] Coronado GD, Schneider JL, Sanchez JJ, Petrik AF, Green B. Reasons for non-response to a direct-mailed FIT kit program: lessons learned from a pragmatic colorectal-cancer screening study in a federally sponsored health center. Transl Behav Med. 2015 Mar;5(1):60-7. doi: 10.1007/s13142-014-0276-x. PMID 25729454
- [Background] Coronado GD, Burdick T, Petrik A, Kapka T, Retecki S, Green B. Using an Automated Data-driven, EHR-Embedded Program for Mailing FIT kits: Lessons from the STOP CRC Pilot Study. J Gen Pract (Los Angel). 2014 Jan 5;2:1000141. doi: 10.4172/2329-9126.1000141. PMID 25411657
- [Background] Coronado GD, Petrik AF, Spofford M, Talbot J, Do HH, Taylor VM. Clinical perspectives on colorectal cancer screening at Latino-serving federally qualified health centers. Health Educ Behav. 2015 Feb;42(1):26-31. doi: 10.1177/1090198114537061. Epub 2014 Jun 20. PMID 24952378
- [Background] Coronado GD, Retecki S, Schneider J, Taplin SH, Burdick T, Green BB. Recruiting community health centers into pragmatic research: Findings from STOP CRC. Clin Trials. 2016 Apr;13(2):214-22. doi: 10.1177/1740774515608122. Epub 2015 Sep 29. PMID 26419905
- [Background] Johnson KE, Tachibana C, Coronado GD, Dember LM, Glasgow RE, Huang SS, Martin PJ, Richards J, Rosenthal G, Septimus E, Simon GE, Solberg L, Suls J, Thompson E, Larson EB. A guide to research partnerships for pragmatic clinical trials. BMJ. 2014 Dec 1;349:g6826. doi: 10.1136/bmj.g6826. No abstract available. PMID 25446054
- [Background] Coronado GD, Petrik AF, Vollmer WM, Taplin SH, Keast EM, Fields S, Green BB. Effectiveness of a Mailed Colorectal Cancer Screening Outreach Program in Community Health Clinics: The STOP CRC Cluster Randomized Clinical Trial. JAMA Intern Med. 2018 Sep 1;178(9):1174-1181. doi: 10.1001/jamainternmed.2018.3629. PMID 30083752
- [Derived] Coronado GD, Nielson CM, Keast EM, Petrik AF, Suls JM. The influence of multi-morbidities on colorectal cancer screening recommendations and completion. Cancer Causes Control. 2021 May;32(5):555-565. doi: 10.1007/s10552-021-01408-2. Epub 2021 Mar 9. PMID 33687606
- [Derived] Petrik AF, Keast E, Johnson ES, Smith DH, Coronado GD. Development of a multivariable prediction model to identify patients unlikely to complete a colonoscopy following an abnormal FIT test in community clinics. BMC Health Serv Res. 2020 Nov 10;20(1):1028. doi: 10.1186/s12913-020-05883-2. PMID 33172444
- [Derived] Petrik AF, Green B, Schneider J, Miech EJ, Coury J, Retecki S, Coronado GD. Factors Influencing Implementation of a Colorectal Cancer Screening Improvement Program in Community Health Centers: an Applied Use of Configurational Comparative Methods. J Gen Intern Med. 2020 Nov;35(Suppl 2):815-822. doi: 10.1007/s11606-020-06186-2. Epub 2020 Oct 26. PMID 33107003
- [Derived] Schneider JL, Rivelli JS, Gruss I, Petrik AF, Nielson CM, Green BB, Coronado GD. Barriers and Facilitators to Timely Colonoscopy Completion for Safety Net Clinic Patients. Am J Health Behav. 2020 Jul 1;44(4):460-472. doi: 10.5993/AJHB.44.4.8. PMID 32553027
- [Derived] O'Connor EA, Vollmer WM, Petrik AF, Green BB, Coronado GD. Moderators of the effectiveness of an intervention to increase colorectal cancer screening through mailed fecal immunochemical test kits: results from a pragmatic randomized trial. Trials. 2020 Jan 15;21(1):91. doi: 10.1186/s13063-019-4027-7. PMID 31941527
- [Derived] Thompson JH, Schneider JL, Rivelli JS, Petrik AF, Vollmer WM, Fuoco MJ, Coronado GD. A Survey of Provider Attitudes, Beliefs, and Perceived Barriers Regarding a Centralized Direct-Mail Colorectal Cancer Screening Approach at Community Health Centers. J Prim Care Community Health. 2019 Jan-Dec;10:2150132719890950. doi: 10.1177/2150132719890950. PMID 31779517
- [Derived] Green BB, Vollmer WM, Keast E, Petrik AF, Coronado GD. Challenges in assessing population reach in a pragmatic trial. Prev Med Rep. 2019 May 29;15:100910. doi: 10.1016/j.pmedr.2019.100910. eCollection 2019 Sep. PMID 31198661
- [Derived] Meenan RT, Coronado GD, Petrik A, Green BB. A cost-effectiveness analysis of a colorectal cancer screening program in safety net clinics. Prev Med. 2019 Mar;120:119-125. doi: 10.1016/j.ypmed.2019.01.014. Epub 2019 Jan 24. PMID 30685318
- [Derived] Nielson CM, Rivelli JS, Fuoco MJ, Gawlik VR, Jimenez R, Petrik AF, Coronado GD. Effectiveness of automated and live phone reminders after mailed-FIT outreach in a pilot randomized trial. Prev Med Rep. 2018 Oct 17;12:210-213. doi: 10.1016/j.pmedr.2018.10.012. eCollection 2018 Dec. PMID 30364785
- [Derived] Coronado GD, Rivelli JS, Fuoco MJ, Vollmer WM, Petrik AF, Keast E, Barker S, Topalanchik E, Jimenez R. Effect of Reminding Patients to Complete Fecal Immunochemical Testing: A Comparative Effectiveness Study of Automated and Live Approaches. J Gen Intern Med. 2018 Jan;33(1):72-78. doi: 10.1007/s11606-017-4184-x. Epub 2017 Oct 10. PMID 29019046
- [Derived] Petrik AF, Le T, Keast E, Rivelli J, Bigler K, Green B, Vollmer WM, Coronado G. Predictors of Colorectal Cancer Screening Prior to Implementation of a Large Pragmatic Trial in Federally Qualified Health Centers. J Community Health. 2018 Feb;43(1):128-136. doi: 10.1007/s10900-017-0395-7. PMID 28744716
- [Derived] Coury J, Schneider JL, Rivelli JS, Petrik AF, Seibel E, D'Agostini B, Taplin SH, Green BB, Coronado GD. Applying the Plan-Do-Study-Act (PDSA) approach to a large pragmatic study involving safety net clinics. BMC Health Serv Res. 2017 Jun 19;17(1):411. doi: 10.1186/s12913-017-2364-3. PMID 28629348
- [Derived] Petrik AF, Green BB, Vollmer WM, Le T, Bachman B, Keast E, Rivelli J, Coronado GD. The validation of electronic health records in accurately identifying patients eligible for colorectal cancer screening in safety net clinics. Fam Pract. 2016 Dec;33(6):639-643. doi: 10.1093/fampra/cmw065. Epub 2016 Jul 28. PMID 27471224
- [Derived] Johnson KE, Neta G, Dember LM, Coronado GD, Suls J, Chambers DA, Rundell S, Smith DH, Liu B, Taplin S, Stoney CM, Farrell MM, Glasgow RE. Use of PRECIS ratings in the National Institutes of Health (NIH) Health Care Systems Research Collaboratory. Trials. 2016 Jan 16;17:32. doi: 10.1186/s13063-016-1158-y. PMID 26772801

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This cluster randomized pragmatic clinical trial was conducted in 26 federally qualified health center clinics, representing 8 health centers in Oregon & California, randomized to intervention (n = 13) or usual care (n = 13). All participants were overdue for colorectal cancer (CRC) screening at some point during accrual interval 2.4.2014-2.3.2015.
Pre-assignment Details: There were 62,155 participants enrolled in the entire study, but 41,193 in the primary analysis.
Units Other Than Participants: Clinics
Groups:
- Usual Care: Usual care clinics continued their standard processes for CRC screening, which typically consisted of providing information and ordering tests during routine clinical encounters. Usual Care clinics were offered training and intervention materials in August 2015.
- Intervention: The intervention consisted of mailed FIT kits, a customized electronic health record (EHR) process and training to support its use.
Period: Overall Study
Arm/Group | Usual Care | Intervention
Started | 20059; 13 Clinics (20059 patients were analyzed in 13 clinics.) | 21134; 13 Clinics (21134 patients were analyzed in 13 clinics.)
Completed | 20059; 13 Clinics (20059 patients were analyzed in 13 clinics.) | 21134; 13 Clinics (21134 patients were analyzed in 13 clinics.)
Not Completed | 0; 0 Clinics | 0; 0 Clinics

BASELINE CHARACTERISTICS:
Population: The baseline analysis was conducted at the clinic level
Units Other Than Participants: Clinics
Groups:
- Usual Care: Usual care clinics continued their standard processes for CRC screening, which typically consisted of providing information and ordering tests during routine clinical encounters
- Total: Total of all reporting groups
Arm/Group | Usual Care | Intervention | Total
Number analyzed (Participants) | 20059 | 21134 | 41193
Number analyzed (Clinics) | 13 | 13 | 26
Age, Customized [Median (Full Range); unit: percentage of participants] — Reported range reflects the range of clinic proportions.
  percentage of participants
    Participants aged 50-64 | 84 [73 to 88] | 80 [73 to 86] | 81 [73 to 88]
    Participants aged 65-75 | 16 [12 to 27] | 20 [14 to 27] | 19 [12 to 27]
Sex/Gender, Customized [Median (Full Range); unit: percentage of participants] — Reported range reflects the range of clinic proportions.
  percentage of participants
    Female | 55 [49 to 65] | 56 [43 to 62] | 56 [43 to 65]
    Male | 45 [35 to 51] | 44 [38 to 57] | 44 [35 to 57]
Race/Ethnicity, Customized [Median (Full Range); unit: percentage of participants] — Data represent the proportion of Hispanic study participants across the individual clinics. Reported range reflects the range of clinic proportions.
  percentage of participants
    Hispanic | 15 [2 to 36] | 8 [1 to 33] | 11 [1 to 36]
Race/Ethnicity, Customized [Median (Full Range); unit: percentage of participants] — Data represent the proportion of study participants by race (categories: white and non-white, other) across the individual clinics. Reported range reflects the range of clinic proportions.
  percentage of participants
    White | 91 [67 to 96] | 93 [50 to 97] | 92 [50 to 97]
    Non-White, other | 5 [2 to 28] | 3 [1 to 40] | 4 [1 to 40]
Region of Enrollment [Number; unit: Clinics]
  United States | 13 | 13 | 26
Language [Median (Full Range); unit: percentage of participants] — Data represent the proportion of study participants by preferred language across the individual clinics. Reported range reflects the range of clinic proportions.
  percentage of participants
    English | 86 [53 to 99] | 90 [41 to 99] | 87 [41 to 99]
    Spanish | 12 [1 to 31] | 4 [0 to 26] | 8 [0 to 31]
    Other | 1 [0 to 18] | 0 [0 to 48] | 1 [0 to 48]
Insurance Status [Median (Full Range); unit: percentage of participants] — Data represent the proportion of study participants by Insurance status across the individual clinics. Reported range reflects the range of clinic proportions.
  percentage of participants
    Medicaid | 35 [25 to 54] | 36 [20 to 51] | 35 [20 to 54]
    Medicare | 23 [15 to 36] | 24 [20 to 37] | 23 [15 to 37]
    Uninsured | 27 [2 to 38] | 26 [3 to 40] | 26 [2 to 40]
    Commercial | 11 [1 to 39] | 10 [1 to 49] | 11 [1 to 49]
Federal Poverty Level [Median (Full Range); unit: percentage of participants] — Data represent the proportion of study participants by federal poverty stratification across the individual clinics. Reported range reflects the range of clinic proportions.
  * <100 represents a household income below the federal poverty level
  * 100-150 represents a household income between 100-150% of the federal poverty level, and so on
  percentage of participants
    <100 percent | 45 [19 to 64] | 47 [13 to 61] | 46 [13 to 64]
    100-150 percent | 18 [14 to 24] | 19 [6 to 31] | 19 [6 to 31]
    151-200 percent | 9 [5 to 13] | 9 [2 to 14] | 9 [2 to 14]
    ≥201percent | 10 [2 to 36] | 10 [3 to 26] | 10 [2 to 36]
    Unknown | 21 [1 to 36] | 17 [3 to 76] | 17 [1 to 76]
Physician Visits in past year [Median (Full Range); unit: percentage of participants] — Data represent the proportion of study participants by number of physician visits in past year across the individual clinics. Reported range reflects the range of clinic proportions.
  percentage of participants
    1 visit | 34 [23 to 44] | 29 [21 to 48] | 33 [21 to 48]
    2-5 visits | 45 [41 to 49] | 46 [40 to 55] | 45 [40 to 55]
    ≥6 visits | 19 [10 to 31] | 19 [9 to 33] | 19 [9 to 33]
% Ever had FIT screening [Median (Full Range); unit: percentage of participants] — Data represent the portion of study participants who have ever had FIT screening across the individual clinics. Reported range reflects the range of clinic proportions.
  percentage of participants | 18 [8 to 39] | 18 [8 to 53] | 18 [8 to 53]
% with Diabetes (ever) [Median (Full Range); unit: percentage of participants] — Data represent the portion of study participants with diabetes diagnosis across the individual clinics. Reported range reflects the range of clinic proportions.
  percentage of participants | 24 [14 to 30] | 22 [13 to 29] | 22 [13 to 30]
% with Flu Shot in past year [Median (Full Range); unit: percentage of participants] — Data represent the portion of study participants with flu shot in the past year across the individual clinics. Reported range reflects the range of clinic proportions.
  percentage of participants | 28 [10 to 40] | 29 [13 to 37] | 29 [10 to 40]
Proportion of Females with Mammogram in past 2 years [Median (Full Range); unit: percentage of participants] — Data represent the proportion of female study participants with a mammogram in the past 2 years across the individual clinics. Reported range reflects the range of clinic proportions. *The percentages are based only on women in the 26 clinics. These data represent the median proportion of women in a clinic with a mammogram. Population: This baseline measure was only assessed in females.
  percentage of participants
    number analyzed (Participants) | 11368 | 11626 | 22994
    (all) | 41 [24 to 59] | 39 [16 to 57] | 40 [16 to 59]
Proportion of Females with Papanicolaou screening in past 3 years [Median (Full Range); unit: percentage of participants] — Data represent the proportion of female study participants with papanicolaou screening in past 3 years across the individual clinics. Reported range reflects the range of clinic proportions.
  *The percentages are based only on women in the 26 clinics. These data represent the median proportion of women in a clinic with papanicolaou screening. Population: This baseline measure was only assessed in females.
  percentage of participants
    number analyzed (Participants) | 11368 | 11626 | 22994
    (all) | 42 [31 to 54] | 42 [15 to 60] | 42 [15 to 60]

OUTCOME MEASURES:

1. Primary Outcome: FIT Completion
Description: Binary indication of FIT completion within 12 months or through August 3, 2015 (when usual care clinics received access to study tools). Proportion of completed FIT is represented below with a confidence interval of the difference in completed FIT.
Time Frame: Completed FIT kits sent back within 12 months
Population: Adult, age 50 to 74 years, clinic visit within 12 months of accrual, and due for CRC screening; no EHR evidence of completed FIT in past 11 months, flexible sigmoidoscopy in past 4 years, colonoscopy in past 9 years, an order for FIT in past 6 months or referral for sigmoidoscopy or colonoscopy in past year.
Measure: Least Squares Mean (95% Confidence Interval); unit: Model based percentage of participants
Groups:
- Intervention: The intervention consisted of mailed FIT kits, a customized EHR process and training to support its use.
Arm/Group | Usual Care | Intervention
Number analyzed (Participants) | 20059 | 21134
Model based percentage of participants | 10.4 [8.1 to 12.8] | 13.9 [11.3 to 16.5]
Statistical Analysis 1: Comparison: Usual Care vs Intervention; Test type: Superiority — To assess effectiveness, we fit generalized estimating equations (GEE) with a logistic link to model patient-level data. We weighted patient data so that each clinic's data had an equal weight. Models were adjusted for age, sex, and health center. They used robust variance estimators and independent correlation structures. We specified clinic as a clustering variable to account for intraclinic correlation; the intraclinic correlation coefficient was 0.05 after model covariates adjustment; p = .05, Generalized Estimating Equations (GEE) — We report effectiveness as the absolute difference between intervention and usual care clinics in adjusted probabilities calculated using mean values for all covariates;; Reported P values based on the corresponding adjusted odds ratio and account for reduced degrees of freedom owing to clustering; Mean Difference (Final Values) = 3.4, 95% CI 2-sided [.1 to 6.8]

2. Secondary Outcome: Any CRC Screening
Description: Binary indication of any CRC screening (fecal test, sigmoidoscopy, or colonoscopy) during the evaluation interval.
Time Frame: Any CRC screening complete within 12 months
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage completed any CRC screening
Arm/Group | Usual Care | Intervention
Number analyzed (Participants) | 20059 | 21134
Percentage completed any CRC screening | 14.5 [12.3 to 16.7] | 18.3 [15.8 to 20.7]
Statistical Analysis 1: Comparison: Usual Care vs Intervention; Test type: Other — To assess effectiveness, we fit generalized estimating equations (GEE) with a logistic link to model patient-level data. We weighted patient data so that each clinic's data had an equal weight. Models were adjusted for age, sex, and health center. They used robust variance estimators and independent correlation structures. We specified clinic as a clustering variable to account for intraclinic correlation; the intraclass correlation coefficient was 0.05 after covariable adjustment; p = .02, Generalized Estimating Equations (GEE) — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 3.8, 95% CI 2-sided [.6 to 7]

ADVERSE EVENTS:
Time Frame: 2.4.2014-8.4.2018, 4.5 years
Description: As our intervention mailed FIT kits to eligible patients (and our primary outcome was completion of FIT), we did not have a systematic way of capturing Severe Adverse Events. Nevertheless, we agreed to document and report to our Data Safety Monitoring Board any Severe Adverse Events we learned about anecdotally from participating clinics, of which there were none.
Groups:
- Usual Care: Usual care clinics continued their standard processes for CRC screening, which typically consisted of providing information and ordering tests during routine clinical encounters. Usual Care clinics were offered training and intervention materials in August 2015, and therefore patients were followed through the end of the study.
- Intervention: The intervention consisted of mailed FIT kits, a customized EHR process and training to support its use. All patients were followed through the end of the study.
Arm/Group | Usual Care | Intervention
All-Cause Mortality (participants affected / at risk) | 0/20059 | 0/21134
Serious Adverse Events (participants affected / at risk) | 0/20059 | 0/21134
Other Adverse Events (participants affected / at risk) | 0/20059 | 0/21134

LIMITATIONS AND CAVEATS:
* FIT samples were not processed if missing collection dates
* under-capture of colonoscopy
* screening/diagnostic colonoscopy indistinguishable
* mailed an introduction letter and having a FIT order served as proxy for having been mailed a FIT.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No